CLINICAL TRIAL: NCT07197905
Title: Restoring Iron Deficiency to Expand Blood Volume and Improve POTS
Brief Title: Restoring Iron Deficiency in POTS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Dysautonomia International (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor of Medicine and Pharmacology, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 250671
Record Dates: First submitted 2025-09-26; First posted 2025-09-30 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: POTS - Postural Orthostatic Tachycardia Syndrome
Keywords: Postural Tachycardia Syndrome; Iron Deficiency
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Iron Deficiencies

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intravenous Iron Infusion (Experimental): The Intravenous iron infusion will be administered according to standard clinical care.
  Interventions: Drug: Intravenous iron

INTERVENTIONS:
Drug: Intravenous iron — The Intravenous iron infusion will be administered according to standard clinical care. The provider will choose the dosage and formulation of IV iron.

SUMMARY:
People with postural orthostatic tachycardia syndrome (POTS) often have low red blood cell volumes and low ferritin in their blood (a marker of iron storage in the body). The purpose of this pilot study is to investigate whether giving iron to people with POTS who have low ferritin levels will increase the red blood cell volume and improve POTS symptoms.

DETAILED DESCRIPTION:
This pilot study involves undergoing a physical exam and medical history, answering some questionnaires, and visiting the Vanderbilt Autonomic Dysfunction Center before and 2 months after the iron treatment for bloodwork, blood volume measurements, autonomic function tests, and wearing an activity monitor.

ELIGIBILITY:
Inclusion Criteria

* Age 18-45 years old.
* Diagnosis of POTS, defined by a sustained heart rate increase of at least 30 bpm within 10 min of standing or head-up tilt (or absolute upright heart rate >120 bpm), in the absence of orthostatic hypotension, and with at least 3 months of symptoms of orthostatic intolerance.
* Absence of other diseases or medications that can explain orthostatic tachycardia or symptoms.
* Serum ferritin <50 ng/ml.
* Patients on fludrocortisone will be allowed to participate as long as they have been on the same dose for at least one month before enrollment and continue on the same dose throughout the study.

Exclusion Criteria

* Unable or unwilling to provide consent.
* Pregnancy.
* Being chair- or bed-ridden.
* Unable to hold POTS medications during study procedures (i.e., autonomic testing).
* History of active bleeding (other than menstruation).
* History of hypersensitivity to any iron preparation of recent (within 6 months) treatment with any IV iron preparation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Orthostatic tachycardia | Orthostatic tachycardia will be assessed before iron infusion (Visit 1) and after 2 months of treatment (Visit 2)
  Orthostatic tachycardia, defined as the difference between upright and supine heart rates, will be assessed during a 10-minute head-up tilt test.

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Autonomic Dysfunction Center/ Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No